CLINICAL TRIAL: NCT01169831
Title: Regulation of Endothelial Progenitor Cells by Short-Term Exercise
Acronym: EPC-Ex
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Baltimore VA Medical Center (U.S. Federal Agency)
Collaborators: University of Maryland, Baltimore (Other); University of Maryland, College Park (Other)
Responsible Party: Principal Investigator, Steven J. Prior, Ph.D., Assistant Professor, University of Maryland, Baltimore
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: HP-00045413
Record Dates: First submitted 2010-07-23; First posted 2010-07-26 (Estimated); Last update posted 2024-08-22 (Actual); Status verified 2024-08

CONDITIONS: Aging; Exercise; Cardiovascular Disease
MeSH Terms: conditions — Motor Activity; Cardiovascular Diseases | interventions — Exercise

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Sedentary Older Adults (Experimental)
  Interventions: Other: Exercise Training
- Older Endurance Athletes (Experimental)
  Interventions: Other: Exercise Cessation

INTERVENTIONS:
Other: Exercise Training — 2 weeks of daily aerobic exercise training
  Arms: Sedentary Older Adults
Other: Exercise Cessation — Stopping all exercise for 2 weeks
  Arms: Older Endurance Athletes

SUMMARY:
Endothelial Progenitor Cells (EPCs) are circulating cells released from bone marrow which are important for maintaining cardiovascular health. The prevalence of cardiovascular disease in older adults is associated with reduced circulating EPC numbers. Studies have shown reduced EPC number and function in old vs. young individuals, and endurance exercise training increases EPC number and function in young adults. Oxidative stress adversely affects endothelial cells and preliminary evidence indicates that oxidative stress negatively affects EPC function. Conversely, regular exercise reduces markers of oxidative stress and may enhance EPC function in older adults. The investigators hypothesize that older endurance-trained athletes and matched sedentary individuals will have markedly divergent EPC function and that altering the physical activity levels of both groups will move them to intermediate points between these two extremes. The investigators also propose that the investigators can "mimic" the effect of exercise training on EPC function in cell culture by altering intracellular levels of a key enzyme and a signaling molecule which the investigators have shown to regulate EPC function with respect to exercise training in young individuals.

ELIGIBILITY:
Inclusion Criteria:

* 50-80 years of age, BMI = 18-35 kg/m2, non-smoking, women must be postmenopausal

Exclusion Criteria:

* history of cardiovascular/cerebrovascular disease, diabetes, cancer, renal, liver disease, HIV; uncontrolled hyperlipidemia/hypertension

Ages: 50 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2011-07; Primary Completion 2014-11 (Actual); Study Completion 2024-07-31 (Actual)

PRIMARY OUTCOMES:
Baseline Endothelial progenitor cell number | Day 1
Final Endothelial Progenitor Cell Number | Day 15

SECONDARY OUTCOMES:
Baseline Endothelial Reactivity | Day 1
Final Endothelial Reactivity | Day 15

CONTACTS AND LOCATIONS:
Overall Officials: Steven J Prior, Ph.D., Principal Investigator — University of Maryland, Baltimore
Locations (1):
- University of Maryland, Baltimore & Baltimore VA Medical Center, Baltimore, Maryland, United States